CLINICAL TRIAL: NCT00958243
Title: A Phase II, Multicenter, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Immunogenicity, Safety and Tolerability of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in a Healthy Pediatric Population
Brief Title: A Clinical Trial of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in a Healthy Pediatric Population in the USA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-CAL-09-62
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- CSL425 (7.5 mcg) (Experimental): 7.5 mcg of hemagglutinin antigen per dose
  Interventions: Biological: CSL's 2009 H1N1 Influenza Vaccine (CSL425)
- CSL425 (15 mcg) (Experimental): 15 mcg of hemagglutinin antigen per dose
  Interventions: Biological: CSL's 2009 H1N1 Influenza Vaccine (CSL425)

INTERVENTIONS:
Biological: CSL's 2009 H1N1 Influenza Vaccine (CSL425) — 0.5 mL intramuscular injection on Day 0 and Day 21
  Arms: CSL425 (15 mcg)
Biological: CSL's 2009 H1N1 Influenza Vaccine (CSL425) — 0.25 mL intramuscular injection on Day 0 and Day 21
  Arms: CSL425 (7.5 mcg)
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety profile of CSL425 (CSL's 2009 H1N1 influenza vaccine) in a healthy pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >= 6 months to < 9 years at the time of the first study vaccination.
* For children < 3 years of age at the time of first vaccination, born at or after 36 weeks gestation.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza virus vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Study Vaccine

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 473 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (13):
- United States (13):
  - Chandler, Arizona
  - Melbourne, Florida
  - Bardstown, Kentucky
  - Metairie, Louisiana
  - Omaha, Nebraska
  - Austintown, Ohio
  - Cincinnati, Ohio
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Murray, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cohort A: Placebo, Aged 6 months to less than 3 years
- CSL425 (7.5 mcg) Cohort A: 7.5 mcg of hemagglutinin antigen per dose, Aged 6 months to less than 3 years
- CSL425 (15 mcg) Cohort A: 15 mcg of hemagglutinin antigen per dose, Aged 6 months to less than 3 years
- Placebo Cohort B: Placebo, Aged 3 years to less than 9 years
- CSL425 (7.5 mcg) Cohort B: 7.5 mcg of hemagglutinin antigen per dose, Aged 3 years to less than 9 years
- CSL425 (15 mcg) Cohort B: 15 mcg of hemagglutinin antigen per dose, Aged 3 years to less than 9 years
Period: Overall Study
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Started | 26 | 105 | 96 | 28 | 109 | 109
Completed | 24 | 99 | 82 | 25 | 100 | 99
Not Completed | 2 | 6 | 14 | 3 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1 | 1 | 5
Not completed — Lost to Follow-up | 2 | 5 | 11 | 2 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B | Total
Number analyzed (Participants) | 26 | 105 | 96 | 28 | 109 | 109 | 473
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 105 | 96 | 28 | 109 | 109 | 473
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.87 (0.77) | 1.73 (0.72) | 1.85 (0.66) | 5.90 (1.71) | 5.94 (1.71) | 5.91 (1.70) | 3.93 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 57 | 44 | 13 | 53 | 50 | 228
  Male | 15 | 48 | 52 | 15 | 56 | 59 | 245
Region of Enrollment [Number; unit: participants]
  United States | 26 | 105 | 96 | 28 | 109 | 109 | 473

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate 21 Days After First Study Vaccination
Description: Seroconversion rate: the percentage of participants achieving seroconversion in HI antibody titer. Seroconversion is defined as participants with a pre-vaccination titer of less than 1:10 achieving a post-vaccination HI antibody titer of 1:40 or more; or participants with a pre-vaccination HI titer of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titer.
Time Frame: 21 days after the first study vaccination
Population: The Evaluable Population (for the first vaccination) comprised all randomized participants who received the first study vaccine; provided both pre- and post-vaccination blood samples; were not excluded from analyses (e.g., the use of a prohibited medication or a laboratory confirmed infection with 2009 H1N1 between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 25 | 102 | 89 | 27 | 104 | 102
Percentage of participants | 4.0 [0.1 to 20.4] | 88.2 [80.4 to 93.8] | 83.1 [73.7 to 90.2] | 3.7 [0.1 to 19.0] | 84.6 [76.2 to 90.9] | 88.2 [80.4 to 93.8]

2. Primary Outcome: Seroconversion Rate 21 Days After Second Study Vaccination
Description: as for outcome 1
Time Frame: 21 days after the second study vaccination
Population: The Evaluable Population (for the second vaccination) comprised all randomized participants who received the second study vaccine; provided both pre- and post-vaccination blood samples; were not excluded from analyses (e.g., the use of a prohibited medication or a laboratory confirmed infection with 2009 H1N1 between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 21 | 90 | 80 | 26 | 98 | 98
Percentage of participants | 28.6 [11.3 to 52.2] | 98.9 [94.0 to 100.0] | 100.0 [95.5 to 100.0] | 15.4 [4.4 to 34.9] | 98.0 [92.8 to 99.8] | 99.0 [94.4 to 100.0]

3. Secondary Outcome: Frequency and Intensity of Solicited Adverse Events (AEs) After the First or Second Study Vaccination, Cohort A
Description: Grade 3 solicited AE definitions: Prevented normal daily activities or required medical intervention for systemic AEs; Cried when limb was moved/spontaneously painful (aged < 3 years) for injection site pain; Size > 30 mm for injection site redness and injection site induration/swelling; Oral temperature > 104.0°F (40.0°C) or axillary temperature > 103.1°F (39.5°C) for fevers.
Time Frame: During the 7 days after each study vaccination
Population: Safety Population comprised all randomized participants who received at least one dose of study vaccine and had provided follow-up safety data.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Cohort A: Placebo
- CSL425 (7.5 mcg) Cohort A: 7.5 mcg of hemagglutinin antigen per dose
- CSL425 (15 mcg) Cohort A: 15 mcg of hemagglutinin antigen per dose
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A
Number analyzed (Participants) | 26 | 105 | 96
Percentage of participants
  Any local solicited adverse event | 42 | 44 | 37
  Any pain | 35 | 33 | 27
  Grade 3 pain | 0 | 0 | 0
  Any redness | 23 | 27 | 19
  Grade 3 redness | 0 | 0 | 0
  Any swelling / induration | 8 | 16 | 6
  Grade 3 swelling / induration | 0 | 0 | 0
  Any systemic solicited adverse event | 58 | 70 | 65
  Any fever | 23 | 25 | 43
  Grade 3 fever | 0 | 3 | 4
  Any nausea / vomiting | 8 | 11 | 15
  Grade 3 nausea / vomiting | 0 | 0 | 0
  Any diarrhea | 39 | 37 | 38
  Grade 3 diarrhea | 0 | 1 | 2
  Any loss of appetite | 12 | 24 | 22
  Grade 3 loss of appetite | 0 | 0 | 1
  Any irritability | 23 | 48 | 34
  Grade 3 irritability | 0 | 1 | 2

4. Secondary Outcome: Duration of Solicited Adverse Events After the First and Second Study Vaccination, Cohort A
Time Frame: During the 7 days after each study vaccination
Population: Safety Population comprised all randomized participants who received at least one dose of study vaccine and had provided follow-up safety data.In Cohort A, Safety Population after the first vaccination are placebo group 26, 7.5 mcg group 105 and 15 mcg group 96; and 25, 101 and 91 respectively after the second vaccination.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A
Number analyzed (Participants) | 26 | 105 | 96
Days
  Any pain after first vaccination | 1.00 (0.000) | 1.52 (0.677) | 1.91 (1.743)
  Any redness after first vaccination | 1.50 (0.577) | 2.20 (1.323) | 2.56 (1.459)
  Any swelling / induration after first vaccination | 1.50 (0.707) | 1.63 (0.957) | 2.00 (1.549)
  Any fever after first vaccination | 3.33 (3.215) | 1.32 (0.557) | 1.29 (0.893)
  Any nausea / vomiting after first vaccination | 1.00 (0.000) | 1.43 (0.535) | 1.11 (0.333)
  Any diarrhea after first vaccination | 1.67 (0.707) | 2.38 (1.996) | 3.95 (4.248)
  Any loss of appetite after first vaccination | 2.00 (NA) — Only one participant reported this AE after the first study vaccination in this group. | 3.13 (2.500) | 2.07 (1.486)
  Any irritability after first vaccination | 6.00 (7.810) | 2.08 (1.412) | 1.97 (1.224)
  Any pain after second vaccination | 1.43 (0.787) | 1.57 (0.676) | 1.23 (0.599)
  Any redness after second vaccination | 2.40 (2.608) | 2.00 (1.240) | 1.63 (0.916)
  Any swelling / induration after second vaccination | 3.00 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 3.00 (2.098) | 2.50 (0.707)
  Any fever after second vaccination | 1.40 (0.894) | 1.40 (0.894) | 2.19 (2.344)
  Any nausea / vomiting after second vaccination | NA (NA) — No participants reported this AE after the second study vaccination in this group. | 1.27 (0.647) | 1.50 (0.837)
  Any diarrhea after second vaccination | 8.00 (9.899) | 1.92 (1.248) | 4.33 (6.754)
  Any loss of appetite after second vaccination | 1.50 (0.707) | 1.75 (1.183) | 3.60 (5.168)
  Any irritability after second vaccination | 1.50 (0.577) | 1.81 (1.001) | 2.86 (4.597)

5. Secondary Outcome: Frequency and Intensity of Solicited Adverse Events After the First or Second Study Vaccination, Cohort B
Description: Grade 3 solicited AE definitions: Prevented normal daily activities or required medical intervention for systemic AEs; Prevented normal daily activities (aged >= 3 years)for injection site pain; Size > 30 mm for injection site redness and injection site induration/swelling; Oral temperature > 104.0°F (40.0°C) or axillary temperature > 103.1°F (39.5°C) for fevers.
Time Frame: During the 7 days after each study vaccination
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Cohort B: Placebo
- CSL425 (7.5 mcg) Cohort B: 7.5 mcg of hemagglutinin antigen per dose
- CSL425 (15 mcg) Cohort B: 15 mcg of hemagglutinin antigen per dose
Arm/Group | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 28 | 107 | 109
Percentage of participants
  Any local solicited adverse event | 43 | 38 | 49
  Any pain | 29 | 34 | 40
  Grade 3 pain | 0 | 0 | 0
  Any redness | 29 | 18 | 26
  Grade 3 redness | 0 | 0 | 0
  Any swelling / induration | 11 | 13 | 17
  Grade 3 swelling / induration | 0 | 0 | 0
  Any systemic solicited adverse event | 46 | 44 | 46
  Any fever | 14 | 19 | 20
  Grade 3 fever | 0 | 0 | 0
  Any nausea / vomiting | 14 | 8 | 13
  Grade 3 nausea / vomiting | 0 | 2 | 1
  Any diarrhea | 21 | 8 | 9
  Grade 3 diarrhea | 0 | 1 | 0
  Any headache | 21 | 17 | 25
  Grade 3 headache | 0 | 1 | 0
  Any malaise | 21 | 27 | 20
  Grade 3 malaise | 4 | 0 | 0
  Any myalgia | 21 | 14 | 22
  Grade 3 myalgia | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants Achieving an Hemagglutination Inhibition (HI) Antibody Titer of 1:40 or More 21 Days After First Study Vaccination
Time Frame: 21 days after the first study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 25 | 102 | 89 | 27 | 104 | 102
Percentage of participants | 8.0 [1.0 to 26.0] | 90.2 [82.7 to 95.2] | 84.3 [75.0 to 91.1] | 25.9 [11.1 to 46.3] | 84.6 [76.2 to 90.9] | 89.2 [81.5 to 94.5]

7. Primary Outcome: Percentage of Participants Achieving an Hemagglutination Inhibition (HI) Antibody Titer of 1:40 or More 21 Days After Second Study Vaccination
Time Frame: 21 days after the second study vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 21 | 90 | 80 | 26 | 98 | 98
Percentage of participants | 28.6 [11.3 to 52.2] | 98.9 [94.0 to 100.0] | 100.0 [95.5 to 100.0] | 34.6 [17.2 to 55.7] | 98.0 [92.8 to 99.8] | 100.0 [96.3 to 100.0]

8. Secondary Outcome: Duration of Solicited Adverse Events After the First and Second Study Vaccination, Cohort B
Time Frame: During the 7 days after each study vaccination
Population: Safety Population comprised all randomized participants who received at least one dose of study vaccine and had provided follow-up safety data. In Cohort B, Safety Population after the first vaccination are placebo group 28, 7.5 mcg group 107 and 15 mcg group 109; and 27, 105 and 103 respectively after the second vaccination.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 28 | 107 | 109
Days
  Any pain after first vaccination | 1.33 (0.516) | 1.63 (1.066) | 1.46 (0.691)
  Any redness after first vaccination | 2.29 (1.254) | 2.17 (1.339) | 2.24 (1.809)
  Any swelling / induration after first vaccination | 2.00 (1.732) | 1.80 (0.632) | 1.79 (0.975)
  Any fever after first vaccination | 1.20 (0.447) | 1.12 (0.332) | 1.56 (0.856)
  Any nausea / vomiting after first vaccination | 1.00 (0.000) | 1.25 (0.500) | 1.00 (0.000)
  Any diarrhea after first vaccination | 1.13 (0.354) | 1.00 (0.000) | 1.22 (0.441)
  Any malaise after first vaccination | 1.38 (0.744) | 1.47 (0.964) | 1.60 (0.995)
  Any myalgia after first vaccination | 1.60 (0.548) | 1.42 (0.669) | 1.56 (0.984)
  Any headache after first vaccination | 1.40 (0.894) | 1.15 (0.376) | 1.25 (0.645)
  Any pain after second vaccination | 1.25 (0.500) | 1.56 (0.856) | 1.33 (0.555)
  Any redness after second vaccination | 2.00 (0.000) | 1.67 (0.516) | 1.60 (0.699)
  Any swelling / induration after second vaccination | 2.00 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 1.17 (0.408) | 1.63 (0.744)
  Any fever after second vaccination | 1.00 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 1.40 (0.548) | 1.57 (1.134)
  Any nausea / vomiting after second vaccination | 1.00 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 1.25 (0.500) | 1.17 (0.408)
  Any diarrhea after second vaccination | 1 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 1.00 (0.000) | 1.00 (0.000)
  Any malaise after second vaccination | 1.50 (0.707) | 1.75 (0.754) | 1.83 (1.467)
  Any myalgia after second vaccination | 1.00 (NA) — Only one participant reported this AE after the second study vaccination in this group. | 1.38 (0.518) | 1.42 (0.669)
  Any headache after second vaccination | 1.50 (0.707) | 1.38 (0.518) | 1.29 (0.488)

9. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAE) After the First or Second Vaccination
Description: UAE grading:
  Grade 1: Symptoms were easily tolerated and did not interfere with daily activities.
  Grade 2: Enough discomfort to cause some interference with daily activities. Grade 3: Symptoms that prevented normal, everyday activities.
Time Frame: During the 21 days after each vaccination
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 26 | 105 | 96 | 28 | 107 | 109
Percentage of participants
  Proportion of participants with at least one UAE | 69 | 52 | 55 | 50 | 49 | 41
  Proportion of participants reported Grade 1 UAE | 31 | 26 | 22 | 14 | 23 | 19
  Proportion of participants reported Grade 2 UAE | 39 | 22 | 27 | 25 | 21 | 17
  Proportion of participants reported Grade 3 UAE | 0 | 5 | 6 | 11 | 5 | 6

10. Secondary Outcome: Incidence of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and New Onset of Chronic Illness (NOCIs)
Description: A NOCI was defined as the diagnosis of a new medical condition that was chronic in nature, including those potentially controllable by medication (e.g., diabetes, asthma).
Time Frame: Up to 180 days after the last vaccination
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Number analyzed (Participants) | 26 | 105 | 96 | 28 | 107 | 109
Percentage of participants
  Proportion of participants with at least one SAE | 0 | 2 | 3 | 0 | 0 | 0
  Proportion of participants with related SAE | 0 | 0 | 0 | 0 | 0 | 0
  Proportion of participants with at least one AESI | 0 | 0 | 0 | 0 | 0 | 0
  Proportion of participants with related AESI | 0 | 0 | 0 | 0 | 0 | 0
  Proportion of participants with at least one NOCI | 0 | 0 | 1 | 0 | 1 | 0
  Proportion of participants with related NOCI | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 180 days after the last study vaccination for SAEs. 21 days after each study vaccination for unsolicited adverse events.
Description: Other adverse events presented are unsolicited adverse events 21 days after either study vaccination.
Arm/Group | Placebo Cohort A | CSL425 (7.5 mcg) Cohort A | CSL425 (15 mcg) Cohort A | Placebo Cohort B | CSL425 (7.5 mcg) Cohort B | CSL425 (15 mcg) Cohort B
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/105 | 3/96 | 0/28 | 0/107 | 0/109
Other Adverse Events (participants affected / at risk) | 25/26 | 58/105 | 82/96 | 22/28 | 70/107 | 49/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort A (N=26) | CSL425 (7.5 mcg) Cohort A (N=105) | CSL425 (15 mcg) Cohort A (N=96) | Placebo Cohort B (N=28) | CSL425 (7.5 mcg) Cohort B (N=107) | CSL425 (15 mcg) Cohort B (N=109)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort A (N=26) | CSL425 (7.5 mcg) Cohort A (N=105) | CSL425 (15 mcg) Cohort A (N=96) | Placebo Cohort B (N=28) | CSL425 (7.5 mcg) Cohort B (N=107) | CSL425 (15 mcg) Cohort B (N=109)
Ear infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 17 (19) | 14 (17) | 3 (3) | 6 (8) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 9 (11) | 17 (21) | 3 (3) | 21 (22) | 15 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 11 (12) | 1 (1) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (7) | 0 (0) | 7 (7) | 2 (2)
Teething (Gastrointestinal disorders) | 1 (1) | 5 (7) | 7 (10) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (5) | 2 (2) | 7 (7) | 2 (2)
Pyrexia (General disorders) | 5 (6) | 8 (8) | 14 (15) | 6 (9) | 15 (17) | 10 (11)
Irritability (General disorders) | 0 (0) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 3 (5)
Malaise (General disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less